CLINICAL TRIAL: NCT04503837
Title: A Randomized Control Trial to Evaluate the Effectiveness of Personalized Mobile Phone Video Recording in Addition to Standard Care Compared to Standard Care Alone in Improving Inhaler Technique Among Patients With Asthma. (RECORD)
Brief Title: Personalized Mobile Phone Video Recording to Improve Inhaler Techniques in Asthma Patients.
Acronym: RECORD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Penang Hospital, Malaysia (Other Government)
Responsible Party: Principal Investigator, Choon Seong Ang, Research Physician, Clinical Research Centre, Penang Hospital, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HPP/CTP/RECORD/01
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Asthma
Keywords: inhaler technique; compliance
MeSH Terms: conditions — Asthma; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All outcome assessment - inhaler technique assessment and asthma control questionnaire will be administered by a blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Personalized Mobile Phone Video Recording in addition to Standard care
  Interventions: Procedure: Personalized Mobile Phone Video Recording
- Control (No Intervention): Standard care alone

INTERVENTIONS:
Procedure: Personalized Mobile Phone Video Recording — Subjects will be asked to perform inhaler technique while on video recording. The video will be shown to subjects immediately during technique education session and mistakes (if any) will be pointed out to subject.
  Arms: Intervention

SUMMARY:
To investigate the effectiveness of addition of recording video of the patient performing inhaler techniques using mobile phone for discussion with the patient, to standard care inhaler education compared to standard care inhaler education alone, in improving inhaler technique of asthma patients.

DETAILED DESCRIPTION:
This is a single-centre, randomized, controlled, parallel group, assessor-blinded trial to evaluate the effectiveness of Personalized Mobile Phone Video Recording in addition to standard care, compared to standard care alone, in improving inhaler technique among patients with asthma.

Patients are randomised to either Personalized Video Recording with standard clinical practice group (intervention) or to standard clinical practice group (control) in 1:1 ratio.

Subject's inhaler technique assessment is performed by using a standard checklist of steps according to the type of inhaler used by subject.

All inhaler technique assessment and asthma control questionnaire will be administered before the intervention/control treatment by a blinded assessor. Both intervention and control treatment will be administered by the same investigators.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and above
2. Informed consent
3. Established clinical diagnosis of asthma by patient's treating doctor
4. Prescribed with inhalers (any type) for therapeutic indication for at least 3 months

Exclusion Criteria:

1. Unable to converse/understand Malay or English
2. Not able to perform inhalation on his/her own self
3. Using spacer/valved holding chamber in addition to MDI
4. Not able to comply with study procedures in the opinion of investigators
5. More than two different types of inhaler which require different techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Inhaler Technique | 6 months
  Correct inhaler technique (able to do all the steps of inhaler technique, as stipulated in checklist of subject's inhaler)

SECONDARY OUTCOMES:
Asthma Control | 1, 3 and 6 months
  Mean score of Asthma Control Questionnaire (ACQ)
Inhaler Technique | 1 and 3 months
  Correct inhaler technique (able to do all the steps of inhaler technique, as stipulated in checklist of subject's inhaler)
Inhaler Technique Error | 1, 3 and 6 months
  Number of errors committed by patients according to checklist

CONTACTS AND LOCATIONS:
Locations (1):
- Penang General Hospital, George Town, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No